CLINICAL TRIAL: NCT01388569
Title: Immune Counter-Regulation in Melanoma Patients Vaccinated With GM-CSF
Brief Title: Biomarkers in Blood Samples From Patients With Stage IV Melanoma Previously Treated With Sargramostim
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000703098; ECOG-E4697T1
Record Dates: First submitted 2011-07-02; First posted 2011-07-06 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Flow Cytometry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: flow cytometry
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients treated with sargramostim in the laboratory may help doctors learn more about the effects of sargramostim on cells. It may also help doctors understand how patients respond to treatment.

PURPOSE: This research trial studies biomarkers in blood samples from patients with stage IV melanoma previously treated with sargramostim.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To correlate circulating myeloid-derived suppressor cells (MDSC) and Treg frequencies with clinical outcome.

Secondary

* To correlate circulating anti-sargramostim (GM-CSF) antibody levels with clinical outcome.

OUTLINE: Archived peripheral blood mononuclear cells and serum samples are analyzed for circulating myeloid-derived suppressor cells, Treg (CD3+/CD4+/CD25hi/FOXP3+) frequency, and anti-sargramostim (anti-GM-CSF) antibody levels by flow cytometry and anti-GM-CSF neutralizing antibody assay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with melanoma

  * Stage IV disease
  * HLA-A2^+ and A2^+
* Received sargramostim on clinical trial ECOG-4697
* Specimens collected at baseline and either day 43 or day 85 (based on most consistent availability) from long-term survivors and patients with poor survival

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patient enrolled on E4697 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2011-09-28 (Actual); Study Completion 2011-09-28 (Actual)

PRIMARY OUTCOMES:
Overall and disease-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Butterfield, PhD, Principal Investigator — University of Pittsburgh